CLINICAL TRIAL: NCT04844216
Title: Effectiveness and Safety of STYLAGE® L Lidocaïne in the Treatment of Nasolabial Folds
Acronym: NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-A03409-30
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Aging
Keywords: Aging; Hyaluronic acid; Nasolabial fold; Injection; Healthy subjects; Independent evaluators; Prospective; Randomized study; Within-subject; Controlled; Multicenter

STUDY DESIGN:
Intervention Model Description: Within-subject study with treatment of one nasolabial fold with the investigational medical device and treatment of the other nasolabial fold with a comparator (another medical device).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Injectors will be unblinded. All subjects, investigators (in charge of clinical examination, assessment of local tolerance, live and on photograph assessment of nasolabial folds severity), as well as technicians (in charge of photographs and measurement of roughness) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasolabial fold treated with experimental device (Experimental): STYLAGE® L Lidocaine is a hyalorunic acid injectable gel whose intended purpose is the filling of skin depressions on the face by dermal injection.
  Up to 2 mL will be injected at Day 0 on a nasolabial fold and, if required, up to 1 mL could be injected 1 month after on the same nasolabial fold (touch-up).
  Interventions: Device: STYLAGE® L Lidocaine
- Nasolabial fold treated with comparator (Active Comparator): The active comparator is a hyalorunic acid injectable gel whose intended purpose is the filling of mid and/or deep depressions of the skin via mid and/or deep dermal injection.
  Up to 2 mL will be injected at Day 0 on a nasolabial fold and, if required, up to 1 mL could be injected 1 month after on the same nasolabial fold (touch-up).
  Interventions: Device: Active control

INTERVENTIONS:
Device: STYLAGE® L Lidocaine — An injection of maximum 2 mL on one nasolabial fold is planned at Day 0. A touch-up of maximum 1 mL on the same nasolabial fold is possible 1 month after D0 (month 1).
  Other Names: Injection of hyaluronic acid gel
  Arms: Nasolabial fold treated with experimental device
Device: Active control — An injection of maximum 2 mL on one nasolabial fold is planned at Day 0. A touch-up of maximum 1 mL on the same nasolabial fold is possible 1 month after D0 (month 1).
  Other Names: Injection of hyaluronic acid gel
  Arms: Nasolabial fold treated with comparator

SUMMARY:
STYLAGE® L Lidocaine is a CE-marked hyaluronic acid gel intended to fill skin depressions on the face by dermal injection. In this study, 50 healthy subjects between the age of 30 and 65, with moderate to severe nasolabial folds as assessed in live, who have given their informed consent and met all eligibility criteria, will be enrolled. Subjects will randomly receive injection of STYLAGE® L Lidocaine on one nasolabial fold and injection of an active comparator on the other nasolabial fold. A touch-up is possible if required one month after. Subjects will come to a total of 7 visits over a period of 12 months. Variation in severity score of nasolabial folds will be assessed in live and on photographs by independent evaluators. Variation in nasolabial fold depth, global aesthetic improvement, subject satisfaction, pain at injection site and safety will also be assessed.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled versus active treatment, within-subjects study with blinded subjects and evaluators assessing the efficay and safety of STYLAGE® L Lidocaine in the treatment of nasolabial folds. Fifty healthy subjects between the age of 30 and 65, with moderate to severe nasolabial folds attaining either grade 3 on both sides or grade 4 on both sides on the Wrinkle Severity Rating Scale (WSRS) for nasolabial folds as assessed in live, who have given their informed consent and met all eligibility criteria, will be enrolled. Subjects will randomly receive dermal injections consisting in a maximum of 2 mL of STYLAGE® L Lidocaine on one nasolabial fold and a maximum of 2 mL of an active comparator on the other nasolabial fold. A touch-up consisting in the dermal injection of maximum 1 mL of product per nasolabial fold is possible if required one month after. Subjects will be followed up at 1, 3, 6, 9 and 12 months timepoints. Variation in severity score of nasolabial folds will be assessed in live and on photographs by independent blinded evaluators using the validated 5-point Wrinkles Severity Rating Scale (WSRS). Global aesthetic improvement will be assessed using the Global Aesthetic Improvement Scale (GAIS). Variation in nasolabial fold depth will be assessed using Dermatop®. Subject satisfaction, pain at injection site and safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Sex: female or male.
* Age: between 30 and 65 years.
* Subject having given freely and expressly his/her informed consent and data privacy consent.
* Subject with approximate symmetry, moderate to severe Nasolabial Folds (NLFs) attaining either grade 3 on both sides or grade 4 on both sides on the Wrinkle Severity Rating Scale (WSRS) for NLF, as assessed in live.
* Subject with marionette's lines that do not require to be treated according to investigator.
* Subject willing to have photographs of the face taken.
* Subject, psychologically able to understand the study related information and to give a written informed consent.
* Subject agreeing not to receive another aesthetic procedure on the face (e.g., laser, dermabrasion, surgery, deep chemical peeling, surface peel, tensor threads, injection with a filling product) during the whole study.
* Subject affiliated to a health social security system.
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before screening visit and during the whole study.

Exclusion Criteria:

* Pregnant or breastfeeding woman or planning a pregnancy during the study.
* Subject with a tattoo, a scar, moles or anything on the studied zones which might interfere with the evaluation.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or who is in an exclusion period of one.
* For France only: subject having received 4500 euros indemnities for participation in researches involving human beings in France in the 12 previous months, including participation in the present study.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject suffering from untreated epilepsy.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject with a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats and in case of acute rheumatic fever with heart complications.
* Subjects suffering from porphyria.
* Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes is not eligible even if asymptomatic at time of screening visit.
* Subject having history of allergy or anaphylactic shock including hypersensitivity to hyaluronic acid, to gram positive bacterial proteins, to lidocaine, to one of the components of the tested devices or antiseptic solution or amide-type local anaesthetics.
* Subject having history of severe and/or evolutive / unstable / recent allergy.
* Subject predisposed to develop keloids or hypertrophic scarring.
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Subjects with known cardiac conduction disorders.
* Subject having received treatment with a laser, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure below the inferior orbital rim within the past 12 months prior to screening visit.
* Subject having received treatment with a surface peel below the inferior orbital rim within the past 6 months prior to screening visit.
* Subject having received injection with a resorbable filling product (eg, hyaluronic acid, collagen) below the inferior orbital rim within the past 12 months prior to screening visit.
* Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable permanent filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …).
* Subject having received at any time a treatment with tensor threads below the inferior orbital rim.
* Subject who received oral surgery (e.g. tooth extraction, orthodontia or implantation) within 6 weeks prior to screening visit or who plans to undergo any of these procedures during the study.
* Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.
* Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAID) (ibuprofène, naproxène, …), antiplatelet agents, anticoagulants, vitamin C or other substances known to prolong bleeding time (warfarin, , herbal supplements with garlic or ginkgo biloba, …) within 1 week prior to injection visit (V1) and agreeing not to take such treatments within 1 week prior to touch-up visit, or being a chronic user.
* Subject using medication that reduce or inhibit hepatic metabolism (cimetidine, beta-blockers, etc).
* Total injection volume of cross-linked hyaluronic acid >14 mL within 1 year prior to screening visit.
* Subject undergoing a topical treatment on the test area or a systemic treatment:

  * Anti-histamines during the 2 weeks prior to injection visit (V1) and agreeing not to take such treatment within 2 weeks prior to touch-up visit;
  * Immunosuppressors and/or corticoids during the 4 weeks prior to screening visit;
  * Retinoids during the 6 months prior to screening visit.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Mean change in nasolabial fold severity assessed in live | Month 6
  Mean change in nasolabial fold severity from baseline to 6 months after treatment initiation, as assessed by an independent blinded live evaluator using the validated 5-point Wrinkles Severity Rating Scale (WSRS). The Wrinkles Severity Rating Scale is a 5-grade scale (from grade 1 to grade 5) with minimum grade representing a better outcome. Grade 1 corresponds to "Absent", grade 2 to "Mild", grade 3 to "Moderate", grade 4 to "Severe" and grade 5 to "Extreme".

SECONDARY OUTCOMES:
Mean change in nasolabial fold severity assessed in live | Month 1, Month 3, Month 9, Month 12
  Mean WSRS change from baseline to 1, 3, 9 and 12 months after treatment initiation, as assessed by an independent blinded live evaluator using the validated 5-point Wrinkles Severity Rating Scale (WSRS).
Mean change in nasolabial fold severity assessed on photographs | Month 1, Month 3, Month 6, Month 9, Month 12
  Mean WSRS change from baseline to 1, 3, 6, 9 and 12 months after treatment initiation as assessed by a blinded independent evaluator on photographs, using the validated 5-point Wrinkles Severity Rating Scale (WSRS).
Evaluation of WSRS responder rate | Month 1, Month 3, Month 6, Month 9, Month 12
  WSRS responder rates 1, 3, 6, 9 and 12 months after treatment initiation as assessed by a blinded live independent evaluator and a blinded independent evaluator on photographs. A responder is defined as a subject with at least 1-point improvement from baseline on the WSRS.
Evaluation of global aesthetic improvement | Month 1, Month 3, Month 6, Month 9, Month 12
  Mean global aesthetic improvement from 1, 3, 6, 9 and 12 months after treatment initiation by subjects and a blinded live independent evaluator using the Global Aesthetic Improvement Scale (GAIS). The Global Aesthetic Improvement Scale is a 5-score scale (from score 1 to score 5) with minimum scores representing a better outcome. Score 1 corresponds to "Very improved", score 2 to "Much improved", score 3 to "Improved", score 4 to "No change" and score 5 to "Worse".
Evaluation of GAIS responder rate | Month 1, Month 3, Month 6, Month 9, Month 12
  GAIS responder rates 1, 3, 6, 9 and 12 months after treatment initiation as assessed by subjects and a blinded live independent evaluator. A responder is defined as a subject having "Improved", "Much improved" or "Very much improved" score according to GAIS.
Mean change in nasolabial fold depth | Month 1, Month 3, Month 6, Month 9, Month 12
  Mean change in nasolabial fold depth from baseline to 1, 3, 6, 9 and 12 months after treatment initiation using Dermatop®.
Evaluation of subject's satisfaction | Month 1, Month 3, Month 6, Month 9, Month 12
  Evaluation of subject's satisfaction 1, 3, 6, 9 and 12 months after treatment initiation using a questionnaire.
Evaluation of pain during injection | Day 0, Month 1
  Evaluation of pain during injection by subjects on an 11-point numeric rating scale (0 to 10).
Report of adverse events | Up to Month 12
  Product tolerance will be assessed by collection of Injection Site Reactions (ISRs) after each injection session, and Adverse Events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CONVERSET-VIETHEL, MD, Principal Investigator — Cabinet de chirugie de la face et du cou
Locations (2):
- Eurofins Dermscan Pharmascan, Villeurbanne, France
- Eurofins Dermscan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No